CLINICAL TRIAL: NCT06757621
Title: Hypofractionated Postoperative Regional Nodal Irradiation for Patients With Intermediate-risk Breast Cancer: A Multicenter Prospective Randomized Phase III Trial and Cohort Study.
Brief Title: Hypofractionated Postoperative Regional Nodal Irradiation for Patients With Intermediate-risk Breast Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Shulian Wang, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC4876; 24/464-4744
Record Dates: First submitted 2024-12-12; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-10

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypofractionated Postoperative Regional Nodal Irradiation (Experimental)
  Interventions: Radiation: Regional Nodal Irradiation
- Without Hypofractionated Postoperative Regional Nodal Irradiation (No Intervention)

INTERVENTIONS:
Radiation: Regional Nodal Irradiation — Patients will receive chest wall / breast radiation with or without regional nodal irradiation
  Arms: Hypofractionated Postoperative Regional Nodal Irradiation

SUMMARY:
The role of postoperative regional nodal irradiation (RNI) for T1-2N1 intermediate-risk breast cancer is controversial, and there is a lack of class I evidence of a survival benefit from RNI. A number of retrospective studies of breast cancer patient been undertaken to risk stratify, analyse site of recurrence and assess the role of radiotherapy. RNI is currently recommended for patients at high risk of recurrence, but prospective studies in other patients are needed to assess the role of RNI. Two randomised phase III trials have confirmed the safety and efficacy of 15-fraction hypofractionated radiotherapy, while 5-fraction super-hypofractionated radiotherapy to further shorten the course of radiotherapy is a hotspot of current research. The present study aimed to investigate whether RNI improves the outcome of intermediate-risk breast cancer patients; and to assess the efficacy and toxicity of 15-fraction hypofractionated and 5-fraction super-hypofractionated radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. ≥45 years old
2. Receiving breast-conserving surgery or total mastectomy and axillary lymph node dissection or sentinel lymph node biopsy
3. Negative surgical margins
4. Tumor staging： A. patients without neoadjuvant chemotherapy: pT1-2N1M0, axillary lymph node dissection with 1-3 metastatic lymph nodes, at least 1 lymph node with macroscopic metastasis, and a score of 0-2 according to the following risk factors: ≤40 years of age (1 point), tumour located in the inner quadrant (1 point), 2-3 lymph nodes positive in the axilla (1 point), presence of choroidal tumour thrombus (1 point), and restaging according to the 8th edition of the staging criteria (IB-IIA 1 point, and IIB-IIIA 2 points) B. patients without neoadjuvant chemotherapy: pT1-2N1M0, sentinel lymph node biopsy with 1-2 metastatic lymph nodes, at least 1 lymph node with macroscopic metastasis, and a score of 0-2 according to the following risk factors: ≤40 years of age (1 point), tumour located in the inner quadrant (1 point), 2-3 lymph nodes positive in the axilla (1 point), presence of choroidal tumour thrombus (1 point), and restaging according to the 8th edition of the staging criteria (IB-IIA 1 point, and IIB-IIIA 2 points) C. patients with neoadjuvant chemotherapy: cT1-2N1-2M0→ypT0-2N0M0, requiring positive clinical lymph nodes with pathological confirmation, receiving ≥6 cycles of neoadjuvant chemotherapy, and ≥3 sentinel lymph nodes detected for those with simple sentinel lymph node biopsy
5. Signed informed consent

Exclusion Criteria:

1. Distant metastases
2. Metastasis to ipsilateral internal breast, supraclavicular or subclavicular lymph nodes
3. Previous radiotherapy to the chest
4. Bilateral breast cancer
5. Pregnancy, breastfeeding
6. Previous or concurrent other malignancy with tumor-free survival <5 years (but excluding skin cancer with non-malignant melanoma, papillary/follicular thyroid cancer, cervical carcinoma in situ)

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3142 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2029-11-01 (Estimated); Study Completion 2032-11-01 (Estimated)

PRIMARY OUTCOMES:
Disease-Free Survival Rate | through study completion, an average of 10 year

SECONDARY OUTCOMES:
Overall Survival Rate | through study completion, an average of 10 year
  Survival
Locoregional Recurrence Rate | through study completion, an average of 10 year
  Survival
Distant Metastasis Rate | through study completion, an average of 10 year
  Survival
Incidence of acute and late adverse reactions | through study completion, an average of 10 year
  CommonTerminology Criteria for Adverse Events (CTCAE) verson 5.0 and Toxicity Criteria of Radiation Therapy Oncology Group (RTOG) are uesd for assessment. Higher toxicity ratings indicate more severe reactions.
Quality of life Questionnaire (EORTC QLQ-C30) | through study completion, an average of 2 year
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) .For the Functioning Scale and the Overall Quality of Life Scale, higher scores indicate better functioning or quality of life
European Organization for Research and Treatment of Cancer Breast Cancer-Specific Quality-of-Life Questionnaire (QLQ-BR23) | through study completion, an average of 2 year
  for the Symptom Scale/Individual Measures, higher scores indicate more severe symptoms or problems.

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
IPD often includes sensitive personal information about patients. Sharing such data could breach patient confidentiality agreements.